CLINICAL TRIAL: NCT05931666
Title: Comparison of Gong and Kaltenborn Mobilization in Frozen Shoulder
Brief Title: Gong v/s Kaltenborn Mobilization in Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIPHAH/RCRS/REC/Letter-01400
Record Dates: First submitted 2023-06-06; First posted 2023-07-05 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Frozen Shoulder
Keywords: Gong mobilization; Kaltenborn mobilization; Frozen shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gong Mobilization (Experimental): The subject placed in a side-lying position with the affected shoulder joint facing upward. and abducted at about 90 degrees to maintain the humerus vertical position with elbow in a 90-degree position. The therapist use one hand to keep the subject's elbow joint at 90 degrees, his elbow below the subject's elbow joint, and the other hand to press the humerus head from anterior to posterior. Therapist elevate own body, pulling on the articular capsule of the shoulder joint. This gentle pulling sustained for 10- 15 seconds before relaxing for 5 seconds; the whole manoeuver last roughly 2-3 minutes.
  Interventions: Other: Gong Mobilization
- Kaltenborn Mobilization (Experimental): Patient lies supine on the table with the arm abducted approximately to 55⁰. The therapist stands facing the lateral side of upper arm. The scapula is fixed using a towel. The therapist's right hand holds around the patients elbow & forearm from the ventral side. Left hand holds around the humeral head with the thumb ventrally just distal to the acromion & the direction of movement is towards caudal assisted by therapist's body. Also anterior and posterior glides are applied with patient positioned similarly in supine lying to improve mobility at the shoulder joint.
  Interventions: Other: Kaltenborn Mobilization

INTERVENTIONS:
Other: Gong Mobilization — Patients are treated with Gong mobilization protocol along with conventional therapy including ultrasound therapy, hot pack and conventional exercises consisting of codman exercises, ROM exercises and shoulder stabilization exercises.
  Total of 3 sessions per week for 3 consecutive weeks.
  Arms: Gong Mobilization
Other: Kaltenborn Mobilization — Patients are treated with Kaltenborn mobilization protocol along with conventional therapy including ultrasound therapy, hot pack and conventional exercises consisting of codman exercises, ROM exercises and shoulder stabilization exercises.
  Total of 3 sessions per week for 3 consecutive weeks.
  Arms: Kaltenborn Mobilization

SUMMARY:
The aim of this research is to determine the effects of Gong mobilization and Kaltenborn mobilization in patients of frozen shoulder. This is a Randomized clinical trial. The sample size is 40. The subjects are divided in two groups, with 20 subjects in Group A and 20 subjects in Group B. Study duration is of 6 months. Sampling technique applied is Nonprobability Purposive Sampling. Both males and females of aged 40-65 years with Stage-II frozen shoulder are included. Tools used in the study are Visual Analogue Scale (VAS), Goniometer, and SPADI (Shoulder pain and disability index) questionnaire.

DETAILED DESCRIPTION:
Adhesive capsulitis or periarthritis, more commonly termed as frozen shoulder is a pathological process where adhesions are formed across glenohumeral joint causing debilitating pain and movement restrictions. The pathology is categorized as primary, being idiopathic and occur spontaneously without any inciting event, or secondary which occur as a result of some identifiable disorder such as diabetes mellitus (where a cascade of inflammatory reactions, collagen build-up and other extracellular components lead to tendon fibrosis and dysfunction, presenting as diabetic frozen shoulder) or some other inciting event. The incidence of frozen shoulder is evident to be 3-5% in general population while it's up to 20% in diabetic patients. Further it is more evident in females aged 40-60 years. Moreover frozen shoulder is classified into four stages which include Stage-I characterized by painful shoulder at rest and disturbed sleep, lasting up to 3 months; Stage-II termed the "freezing stage" is identified by chronic pain along with restrictions in range of motion (ROM) and last up to 9 months; Stage-III called the "frozen stage" where a considerable reduction in ROM and a rigid end feel is observed and occurs during 9 to 15 months of onset; Stage-IV is "thawing phase" where ROM improves progressively, as frozen shoulder is a self-limiting condition and lasts from 15 to 24 months.

The standard exercise protocol followed for management of frozen shoulder include active and active assisted exercises, Codman exercises, wall and ladder exercises, wand exercises, capsular stretching, and shoulder joint mobilization. The electrotherapeutic modalities employed include ultrasound to resolve inflammation, interferential therapy and transcutaneous electrical nerve stimulation (TENS) for pain control and thermal therapy to relieve pain and improve muscles extensibility.

Manual therapy techniques of mobilization have been proved to be very effective in treating frozen shoulder. The Gong's mobilization technique which combines the concepts of distraction and Maitland, is explained as end range mobilization where an antero-posterior glide is applied in dynamic position of the shoulder joint followed by distraction and performance of the restricted movement. The technique serves to reduce pain and improve range of motion and is significant in producing immediate effects. Kaltenborn mobilization technique depends on concave rule and gives grades of traction which include loosening, tightening and stretching of the soft connective tissues.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral stage-II frozen shoulder.
* Both males and females.
* Subjects within 40- 65 years age.
* Capsular pattern restrictions in ROM (external rotation is more limited than abduction, which is more limited than internal rotation).

Exclusion Criteria:

* Subjects with previous surgery of the shoulder joint.
* Subjects with rotator cuff rupture.
* History of recent fracture or severe trauma to the shoulder.
* Restricted shoulder ROM due to burns or postoperative scars.
* Diagnosed instability or previous history of dislocation
* Systemic inflammatory conditions (e.g. rheumatoid arthritis)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Shoulder pain and disability index | 3rd week
  SPADI was developed to measure the pain and disability associated with shoulder pathology. The SPADI is a self-administered index consisting of 13 items divided into two subscales i.e. pain and disability. A remarkably good internal consistency and high test-retest reliability value was found (ICC for pain=0.989 [95% CI=0.975-0.995]; ICC for disability=0.990 [95% CI=0.988-0.998]

SECONDARY OUTCOMES:
Visual Analogue Scale | 3rd week
  Visual Analogue Rating (VAS) is a self-report of clinical pain intensity. The scale was 10 cm long and anchored by the statements "no pain" (0-4 mm) on the left mild pain (5-44 mm), moderate pain (45-74 mm), and the most intense pain imaginable (75-100 mm) on the right. It is a reliable tool with ICC (95% CI) value 0.97 (0.96-0.98). VAS is considered to have good construct validity i.e. highly correlated with numeric rating scale and verbal rating scale with correlations values 0.941 and 0.878 respectively
Shoulder ranges using Goniometer | 3rd week
  A device used by physical therapists to measure joints' range of motion. During measurement fulcrum will be placed on shoulder joint parallel to sagittal axis for abduction and adduction, frontal axis for flexion and extension and to humeral longitudinal axis in 90o of abduction for internal and external rotations. The intra class correlation coefficients (ICC) validity ranged from 0.945 to 0.973 for the goniometric measurements

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PhD*, Principal Investigator — Riphah College of Rehabilitation and Allied Health Sciences, Riphah International University
Locations (2):
- Pakistan (2):
  - Satellite Specialist Clinic, Rawalpindi, Punjab Province
  - Professional Specialist Rehab Center, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No